CLINICAL TRIAL: NCT00122785
Title: Efficacy of Single Injection of Dexamethasone for Acute Bronchiolitis in Children Younger Than 2 Years Old: A Randomized, Double-Blind, Placebo Controlled Trial
Brief Title: Single Injection of Dexamethasone for Acute Bronchiolitis in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE44243
Record Dates: First submitted 2005-07-18; First posted 2005-07-22 (Estimated); Last update posted 2005-07-29 (Estimated); Status verified 2005-02

CONDITIONS: Bronchiolitis, Viral
Keywords: bronchiolitis; wheezing; dexamethasone; young children
MeSH Terms: conditions — Bronchiolitis, Viral; Bronchiolitis; Respiratory Sounds | interventions — Dexamethasone

INTERVENTIONS:
Drug: dexamethasone

SUMMARY:
The purpose of this study was to determine whether a single intramuscular injection of dexamethasone decreased the duration of symptoms of acute bronchiolitis in young children.

DETAILED DESCRIPTION:
Acute bronchiolitis is an infection of the lower respiratory tract causing inflammation of the small airways, leading to bronchiolar obstruction. Corticosteroids are frequently prescribed as anti-inflammatory drugs. The usefulness of corticosteroids for this disease remains controversial, despite many randomized controlled trials (RCTs). Recently, a meta-analysis and systemic review showed significant improvement in clinical symptoms, length of hospital stay and duration of symptoms in children with this disease after treatment with various regimens of systemic corticosteroids.

Dexamethasone is a long acting corticosteroid with biologic half-life ranging from 36-72 hours. A single dose of dexamethasone has been the standard recommendation for the treatment of croup which has a similar pathophysiology without evidence of adverse effects. Furthermore, there is no previous report of this single dosage form of dexamethasone for the treatment of acute bronchiolitis in young children.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 weeks - 24 months
* Has the first episode of wheezing within 7 days
* Has evidence of viral infection
* Requires hospital admission; criteria for admission include one of the following: age < 3 months; respiratory rate > 60 breaths/minute for age < 12 months or 50 breaths/minute for > or equal to 12 months; oxygen saturation in room air < 95% and apathy or refuses feeding.

Exclusion Criteria:

* Initial admission to intensive care unit
* Initial requirement for endotracheal intubation or mechanical ventilation
* A previous history of intubation
* A known history of asthma or response to the first dose of beta2 agonist nebulization
* A history of prematurity
* A history of bronchopulmonary dysplasia or chronic lung disease
* Underlying congenital heart disease or immunodeficiency
* Receives treatment of any form of corticosteroids within 2 weeks
* Has contraindication to corticosteroid treatment

Ages: 4 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170
Dates: Start 2002-04; Study Completion 2004-09

PRIMARY OUTCOMES:
The time from study entry to respiratory distress resolved, which was defined as the following: respiratory rate score of 0 or 1
wheezing score of 0 or 1
retraction muscle score of 0 or 1
and oxygen saturation greater than or equal to 95% without oxygen

SECONDARY OUTCOMES:
The duration of oxygen therapy
The length of hospital stay
Additional drugs used
Emergency visit and hospital readmission within one month after discharge
Adverse drug events

CONTACTS AND LOCATIONS:
Overall Officials: Jamaree Teeratakulpisarn, M.D., Principal Investigator — Faculty of Medicine, Khon Kaen University, Thailand
Locations (1):
- Srinagarind Hospital, Khon Kaen University and Khon Kaen Hospital, Ministry of Public Health, Khon Kaen, Changwat Khon Kaen, Thailand